CLINICAL TRIAL: NCT00671710
Title: A Phase 1 and 2 Study of Aminolevulinic Acid (ALA) to Enhance Visualization and Resection of Malignant Glial Tumors of the Brain
Brief Title: Study of Aminolevulinic Acid to Enhance Visualization and Resection of Malignant Glial Tumors of the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Advocate Hospital System (Other)
Responsible Party: John Ruge, M.D., Advocate Lutheran General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4079
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2010-06

CONDITIONS: Brain Tumors
Keywords: malignant glial brain tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aminolevulinic Acid — Escalating doses (10mg/kg, 20mg/kg, 30mg/kg) of Aminolevulinic Acid administered orally 3 hours prior to surgery to enhance visualization of malignant brain tumor.
  Other Names: ALA

SUMMARY:
Tumors of the central nervous system are potentially curable. For tumors of comparable histology and grade, resectability is the most important prognostic factor affecting survival particularly in children. However, the infiltrative nature of the malignant cells produces indistinct borders between normal and malignant tissues, and the lack of easily identifiable tumor margins confounds attempts toward total resection. The investigators propose to identify the borders of tumors intraoperatively using protoporphyrin fluorescence of the malignant cells and thereby provide more complete tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* patients must have clinically documented primary brain tumor for which resection is clinically indicated. Anticipated histology at resection should include:anaplastic astrocytoma, astrocytoma malignant NOS,brain stem glioma, ependymoma malignant, glioblastoma, glioblastoma multiforme, gliosarcoma, malignant oligodendroglioma, medulloblastoma, mixed astrocytoma-ependymoma
* prior therapy is not a consideration in protocol entry
* age unrestricted
* ECOG performance status<2(Karnofsky>60%,)
* life expectancy is not a consideration for protocol entry
* patients must have normal organ and marrow function as defined below:
* leukocytes _> 3,000/ml
* absolute neutrophil count _>1,500/ml
* platelets >_100,000/ml
* total bilirubin:within normal institutional limits
* AST (SGOT)/ALT (SGPT) _<2.5 X institutional upper limit of normal
* creatinine:within normal institutional limits or creatinine clearance >_60 ml/min/1.73 m2 for patients with creatinine levels above institutional normal
* women of child-bearing potential and men must agree to use adequate contraception(hormonal or barrier method of birth control;abstinence) prior to study entry and for the duration of study participation.
* ability to understand and the willingness to sign a written informed consent document or have a parent or guardian with the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* prior therapy is not an exclusion criterion
* patients may not be receiving any other investigational agents history of allergic reactions attributed to compounds of similar chemical or biologic composition to aminolevulinic adic (ALA)
* personal or family history of porphyrias
* uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* pregnant women are excluded, breastfeeding should be discontinued if mother is treated with aminolevulinic acid.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Establish safe dose for oral ALA administration. NCI Common Toxicity Criteria will be used to quantify toxicity following ALA administration. | 108 weeks

SECONDARY OUTCOMES:
Compare time-to-progression and survival to that in comparable cases performed without the aid of ALA. Kaplan-Meier plots of survival and TTP will be generated for all study subjects and for patients at the 30 mg/kg dose level alone. | 108 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Ruge, M.D., Principal Investigator — Advocate Lutheran General Hospital
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States